CLINICAL TRIAL: NCT01048970
Title: A Prospective Randomized Trial: Effect of Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA)- Containing Supplement on the Nutritional and Inflammatory Status, Quality of Life, Toxicity and Response Rate to First-line Chemotherapy in Patients With Advanced Lung Cancer
Brief Title: Effect on the Nutritional and Inflammatory Status of Docosahexaenoic Acid (DHA) and Eicosapentaenoic Acid (EPA)- Containing Supplement in Patients With Advanced Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Oscar Arrieta, National Institute of Cancerologia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INCAN/CC/330/09; CA171/CB/558/09 (Other: National Institute of Cancerologia)
Record Dates: First submitted 2010-01-09; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Eicosapentaenoic acid oral supplementation; Weight loss; Toxicity; Body composition; Inflammatory response
MeSH Terms: conditions — Lung Neoplasms; Weight Loss | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Other): Patients will receive nutritional assessment one week prior to treatment until completing two cycles
  Interventions: Other: Nutritional Assessment
- EPA-DHA arm (Experimental): Patients will be randomized to receive two cans/day of EPA and DHA containing oral supplement one week prior to treatment until completing two courses of chemotherapy
  Interventions: Dietary Supplement: EPA-DHA arm

INTERVENTIONS:
Other: Nutritional Assessment — Patients will receive nutritional assessment one week prior to treatment until completing two courses of chemotherapy
  Arms: Control arm
Dietary Supplement: EPA-DHA arm — Patients will be randomized to receive two cans/day of EPA and DHA containing oral supplement one week prior to treatment until completing two courses of chemotherapy
  Arms: EPA-DHA arm

SUMMARY:
Background: A frequent manifestation of advanced lung cancer is malnutrition, timely identification and treatment of which can lead to improved patient quality of life, response rate to chemotherapy and survival. N-3 fatty acids, especially eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), may possess anticachectic properties. This trial compared a protein and energy dense supplement enriched with n-3 fatty acids with nutritional assessment for their effects on weight, lean body mass (LBM), body fat, phase angle, dietary intake, inflammatory response and quality of life in first-line chemotherapy patients with advanced lung cancer.

Methods: Chemonaive patients with stages IIIB and IV of lung cancer are going to receive Paclitaxel and Cisplatin. Patients will be randomized to receive two cans/day of EPA and DHA containing oral supplement or nutritional assessment one week prior to treatment until completing two cycles. Serum levels of Reactive C Protein (RCP), interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-alpha) are going to be measured baseline and after two courses of chemotherapy. Phase angle and body composition will be measured using Bioimpedance analysis (BIA). Quality of life, dietary intake will be assessed with validate questionnaires. All data is going to be collected in a database for further blind analysis. Written informed consent will be collected from all patients.

DETAILED DESCRIPTION:
Background: A frequent manifestation of advanced lung cancer is malnutrition, timely identification and treatment of which can lead to improved patient quality of life, response rate to chemotherapy and survival. N-3 fatty acids, especially eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), may possess anticachectic properties. This trial compared a protein and energy dense supplement enriched with n-3 fatty acids with nutritional assessment for their effects on weight, lean body mass (LBM), body fat, phase angle, dietary intake, inflammatory response and quality of life in first-line chemotherapy patients with advanced lung cancer.

Hypothesis: Lung cancer patients who received EPA and DHA containing oral supplement will have a lower frequency of weight loss, rate of adverse effects to chemotherapy and inflammatory response, improving quality of life, response rate to chemotherapy compared with patients who received nutritional assessment.

Methods: Chemonaive patients with stages IIIB and IV of lung cancer are going to receive Paclitaxel and Cisplatin. Patients will be randomized to receive two cans/day of EPA and DHA containing oral supplement or nutritional assessment one week prior to treatment until completing two cycles. Serum levels of Reactive C Protein (RCP), interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-alpha) are going to be measured baseline and after two courses of chemotherapy. Phase angle and body composition will be measured using Bioimpedance analysis (BIA). Quality of life, dietary intake will be assessed with validate questionnaires. All data is going to be collected in a database for further blind analysis. Written informed consent will be collected from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology diagnosis of stage IIIB or IV lung cancer.
* Patients who will received paclitaxel 175 mg/m2 and cisplatin 75 mg/m2 chemotherapy treatment each 3 weeks.
* ECOG < 2.
* Hepatic, nephrotic and hematology laboratories in normal ranges.

Exclusion Criteria:

* Patients who do not accept to participate.
* Patients who have been received chemotherapy treatment.
* Patients with current nutritional assessment and/or nutritional supplements intake.
* Patients with poor performance status.
* Pregnant or lactating women.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory response | 12 months
Response rate to chemotherapy | 1 year
Quality of life | 1 year
Nutritional status | 1 year

SECONDARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — National Institute of Cancerología
Locations (2):
- Mexico (2):
  - National Institute of Cancerologia, Mexico City, Mexico City
  - National Institute of Cancerología, Mexico City, Mexico City

REFERENCES:
- [Background] Fearon KC, Von Meyenfeldt MF, Moses AG, Van Geenen R, Roy A, Gouma DJ, Giacosa A, Van Gossum A, Bauer J, Barber MD, Aaronson NK, Voss AC, Tisdale MJ. Effect of a protein and energy dense N-3 fatty acid enriched oral supplement on loss of weight and lean tissue in cancer cachexia: a randomised double blind trial. Gut. 2003 Oct;52(10):1479-86. doi: 10.1136/gut.52.10.1479. PMID 12970142
- [Background] Gupta D, Lammersfeld CA, Vashi PG, King J, Dahlk SL, Grutsch JF, Lis CG. Bioelectrical impedance phase angle in clinical practice: implications for prognosis in stage IIIB and IV non-small cell lung cancer. BMC Cancer. 2009 Jan 28;9:37. doi: 10.1186/1471-2407-9-37. PMID 19175932
- [Background] Dewey A, Baughan C, Dean T, Higgins B, Johnson I. Eicosapentaenoic acid (EPA, an omega-3 fatty acid from fish oils) for the treatment of cancer cachexia. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD004597. doi: 10.1002/14651858.CD004597.pub2. PMID 17253515
- [Derived] Sanchez-Lara K, Turcott JG, Juarez-Hernandez E, Nunez-Valencia C, Villanueva G, Guevara P, De la Torre-Vallejo M, Mohar A, Arrieta O. Effects of an oral nutritional supplement containing eicosapentaenoic acid on nutritional and clinical outcomes in patients with advanced non-small cell lung cancer: randomised trial. Clin Nutr. 2014 Dec;33(6):1017-23. doi: 10.1016/j.clnu.2014.03.006. Epub 2014 Apr 4. PMID 24746976